CLINICAL TRIAL: NCT01832311
Title: Protein Profile of Immunoregulatory Factors in Diabetic Cataract
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Danka Grcevic, prof. Danka Grcevic, MD, PhD, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 108-1080229-0142
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Cataract; Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; cataract; cytokines; chemokines; aqueous humor
MeSH Terms: conditions — Cataract; Diabetes Mellitus, Type 2 | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- senile cataract with NSAID (Experimental): 15 non-diabetic patients undergoing phacoemulsification combined with IOL implantation.
  Subgroup receiving topical nonsteroidal anti-inflammatory drug (NSAID) ketorolac.
  Interventions: Drug: Ketorolac
- diabetic cataract with NSAID (Experimental): 17 diabetic patients undergoing phacoemulsification combined with IOL implantation.
  Subgroup receiving topical nonsteroidal anti-inflammatory drug (NSAID) ketorolac.
  Interventions: Drug: Ketorolac
- senile cataract without NSAID (No Intervention): 17 non-diabetic patients undergoing phacoemulsification combined with IOL implantation.
  Subgroup not receiving topical ketorolac.
- diabetic cataract without NSAID (No Intervention): 12 diabetic patients undergoing phacoemulsification combined with IOL implantation.
  Subgroup not receiving topical ketorolac.

INTERVENTIONS:
Drug: Ketorolac — Patients (both non-diabetic and diabetic) were randomized into subgroups receiving topical nonsteroidal anti-inflammatory drug (NSAID) ketorolac 0.5%, dosed 4 times a day, starting 3-7 days before surgery and ending 4-5 weeks after surgery respectively, and into subgroups not receiving NSAID.
  Other Names: Toradol; Acular; Sprix
  Arms: diabetic cataract with NSAID; senile cataract with NSAID

SUMMARY:
The purpose of this study is to compare the levels of several immunoregulatory factors in serums and aqueous humor of type II diabetes cataract patients with those in senile non-diabetic cataract patients since disturbed cytokine and growth factor microenvironment in diabetic eye may contribute to an increased frequency of intraoperative and postoperative intraocular lens surgery complications.

DETAILED DESCRIPTION:
The study compared the levels of several immunoregulatory molecules (vascular endothelial growth factor (VEGF), monocyte chemotactic protein-1 (MCP-1), Fas Ligand (FasL), interleukin-10 (IL-10) and interleukin-17 (IL-17)) in serum and aqueous humor between type 2 diabetes mellitus patients, without clinically evident diabetic retinopathy or diabetic macular edema, and nondiabetic cataract patients.

Investigators also investigated whether concentrations of immunoregulatory molecules significantly correlated with intraoperative and postoperative parameters. Particularly, investigators focused on the development of corneal edema as one of the main causes of low visual acuity in the immediate postoperative period after intraocular lens implantation.

Since disturbed cytokine and growth factor microenvironment in diabetic eye may contribute to an increased frequency of intraoperative and postoperative intraocular lens (IOL) surgery complications, the findings may be relevant for the development of therapeutic strategies aimed to restore protein profile of immunoregulatory factors in parallel to cataract treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing phacoemulsification combined with IOL implantation
* for diabetic group: duration of type 2 diabetes mellitus (T2DM) for 10 to 15 years
* for diabetic group: therapy with oral hypoglycemic agents for glycemic control
* no other ocular (retinal) or systemic diabetic complications of T2DM

Exclusion Criteria:

* patients who had cataract that could result from some other ocular condition, systemic disease (except T2DM for diabetic group) or trauma
* patients with immune disease, local or systemic inflammation which could affect cytokine concentration in serum or aqueous humor (AH)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
serum level of interleukin-10 | 2 hours before the surgery
serum level of monocyte chemotactic protein-1 | 2 hours before the surgery
serum level of interleukin-17 | 2 hours before the surgery
serum level of Fas ligand | 2 hours before the surgery
serum level of vascular endothelial growth factor | 2 hours before the surgery
level of interleukin-10 in aqueous humor | intraoperatively, at the start of the surgical procedure
level of monocyte chemotactic protein-1 in aqueous humor | intraoperatively, at the start of the surgical procedure
level of interleukin-17 in aqueous humor | intraoperatively, at the start of the surgical procedure
level of Fas ligand in aqueous humor | intraoperatively, at the start of the surgical procedure
level of vascular endothelial growth factor in aqueous humor | intraoperatively, at the start of the surgical procedure

SECONDARY OUTCOMES:
degree of corneal edema | preoperatively - 2 hours before the surgery
degree of corneal edema | postoperatively - day 1
degree of corneal edema | postoperatively - day 8
degree of corneal edema | postoperatively - week 3
degree of corneal edema | postoperatively - month 3

CONTACTS AND LOCATIONS:
Overall Officials: Danka Grcevic, prof.,MD,PhD, Principal Investigator — University of Zagreb; Sanja Mitrovic, MD, Principal Investigator — Department of Ophthalmology, General Hospital "Dr. J. Bencevic"
Locations (2):
- Croatia (2):
  - Department of Ophtalmology, General Hospital "Dr. J. Bencevic", Slavonski Brod, Brod-Posavina County
  - Department of Physiology and Immunology, University of Zagreb School of Medicine, Zagreb, City of Zagreb

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Benson WE. Cataract surgery and diabetic retinopathy. Curr Opin Ophthalmol. 1992 Jun;3(3):396-400. doi: 10.1097/00055735-199206000-00015. PMID 10149703
- [Background] Klein BE, Klein R, Moss SE. Prevalence of cataracts in a population-based study of persons with diabetes mellitus. Ophthalmology. 1985 Sep;92(9):1191-6. doi: 10.1016/s0161-6420(85)33877-0. PMID 4058882
- [Background] Nielsen NV, Vinding T. The prevalence of cataract in insulin-dependent and non-insulin-dependent-diabetes mellitus. Acta Ophthalmol (Copenh). 1984 Aug;62(4):595-602. doi: 10.1111/j.1755-3768.1984.tb03972.x. PMID 6385608
- [Background] Hamilton AMP (1996) Epidemiology of Diabetic Retinopathy. In: Hamilton AMP, Ulbig MW, Polkinghorne P (eds) Management of Diabetic Retinopathy. B.M.J. Publishing Group, London, pp. 1-15
- [Background] Obrosova IG, Minchenko AG, Vasupuram R, White L, Abatan OI, Kumagai AK, Frank RN, Stevens MJ. Aldose reductase inhibitor fidarestat prevents retinal oxidative stress and vascular endothelial growth factor overexpression in streptozotocin-diabetic rats. Diabetes. 2003 Mar;52(3):864-71. doi: 10.2337/diabetes.52.3.864. PMID 12606532
- [Background] Pollreisz A, Schmidt-Erfurth U. Diabetic cataract-pathogenesis, epidemiology and treatment. J Ophthalmol. 2010;2010:608751. doi: 10.1155/2010/608751. Epub 2010 Jun 17. PMID 20634936
- [Background] Funatsu H, Yamashita H, Noma H, Mimura T, Yamashita T, Hori S. Increased levels of vascular endothelial growth factor and interleukin-6 in the aqueous humor of diabetics with macular edema. Am J Ophthalmol. 2002 Jan;133(1):70-7. doi: 10.1016/s0002-9394(01)01269-7. PMID 11755841
- [Background] Gverovic Antunica A, Karaman K, Znaor L, Sapunar A, Busko V, Puzovic V. IL-12 concentrations in the aqueous humor and serum of diabetic retinopathy patients. Graefes Arch Clin Exp Ophthalmol. 2012 Jun;250(6):815-21. doi: 10.1007/s00417-011-1905-4. Epub 2012 Jan 8. PMID 22227739
- [Background] Jonas JB, Jonas RA, Neumaier M, Findeisen P. Cytokine concentration in aqueous humor of eyes with diabetic macular edema. Retina. 2012 Nov-Dec;32(10):2150-7. doi: 10.1097/IAE.0b013e3182576d07. PMID 22617833
- [Background] Cheung CM, Vania M, Ang M, Chee SP, Li J. Comparison of aqueous humor cytokine and chemokine levels in diabetic patients with and without retinopathy. Mol Vis. 2012;18:830-7. Epub 2012 Apr 4. PMID 22511846
- [Background] Hernandez C, Segura RM, Fonollosa A, Carrasco E, Francisco G, Simo R. Interleukin-8, monocyte chemoattractant protein-1 and IL-10 in the vitreous fluid of patients with proliferative diabetic retinopathy. Diabet Med. 2005 Jun;22(6):719-22. doi: 10.1111/j.1464-5491.2005.01538.x. PMID 15910622
- [Background] Funatsu H, Yamashita H, Sakata K, Noma H, Mimura T, Suzuki M, Eguchi S, Hori S. Vitreous levels of vascular endothelial growth factor and intercellular adhesion molecule 1 are related to diabetic macular edema. Ophthalmology. 2005 May;112(5):806-16. doi: 10.1016/j.ophtha.2004.11.045. PMID 15878060
- [Background] Stefek M, Karasu C. Eye lens in aging and diabetes: effect of quercetin. Rejuvenation Res. 2011 Oct;14(5):525-34. doi: 10.1089/rej.2011.1170. Epub 2011 Oct 6. PMID 21978083
- [Background] Crandall AS, Zabriskie NA, Patel BC, Burns TA, Mamalis N, Malmquist-Carter LA, Yee R. A comparison of patient comfort during cataract surgery with topical anesthesia versus topical anesthesia and intracameral lidocaine. Ophthalmology. 1999 Jan;106(1):60-6. doi: 10.1016/S0161-6420(99)90007-6. PMID 9917782
- [Background] Altintas AG, Yilmaz E, Anayol MA, Can I. Comparison of corneal edema caused by cataract surgery with different phaco times in diabetic and non-diabetic patients. Ann Ophthalmol (Skokie). 2006 Spring;38(1):61-5. doi: 10.1385/ao:38:1:61. PMID 17200587
- [Background] Amon M, Menapace R, Scheidel W. Results of corneal pachymetry after small-incision hydrogel lens implantation and scleral-step incision poly(methyl methacrylate) lens implantation following phacoemulsification. J Cataract Refract Surg. 1991 Jul;17(4):466-70. doi: 10.1016/s0886-3350(13)80853-x. PMID 1895223
- [Background] Brazitikos PD, Androudi S, Papadopoulos NT, Christen WG, Stangos NT. A-scan quantitative echography of senile cataracts and correlation with phacoemulsification parameters. Curr Eye Res. 2003 Sep;27(3):175-81. doi: 10.1076/ceyr.27.3.175.16051. PMID 14562183
- [Background] Tabandeh H, Wilkins M, Thompson G, Nassiri D, Karim A. Hardness and ultrasonic characteristics of the human crystalline lens. J Cataract Refract Surg. 2000 Jun;26(6):838-41. doi: 10.1016/s0886-3350(00)00305-9. PMID 10889428
- [Background] Oh IK, Kim SW, Oh J, Lee TS, Huh K. Inflammatory and angiogenic factors in the aqueous humor and the relationship to diabetic retinopathy. Curr Eye Res. 2010 Dec;35(12):1116-27. doi: 10.3109/02713683.2010.510257. PMID 21121809
- [Background] Schoenberger SD, Kim SJ, Sheng J, Rezaei KA, Lalezary M, Cherney E. Increased prostaglandin E2 (PGE2) levels in proliferative diabetic retinopathy, and correlation with VEGF and inflammatory cytokines. Invest Ophthalmol Vis Sci. 2012 Aug 27;53(9):5906-11. doi: 10.1167/iovs.12-10410. PMID 22871833
- [Background] Tashimo A, Mitamura Y, Nagai S, Nakamura Y, Ohtsuka K, Mizue Y, Nishihira J. Aqueous levels of macrophage migration inhibitory factor and monocyte chemotactic protein-1 in patients with diabetic retinopathy. Diabet Med. 2004 Dec;21(12):1292-7. doi: 10.1111/j.1464-5491.2004.01334.x. PMID 15569131
- [Background] Mine S, Okada Y, Tanikawa T, Kawahara C, Tabata T, Tanaka Y. Increased expression levels of monocyte CCR2 and monocyte chemoattractant protein-1 in patients with diabetes mellitus. Biochem Biophys Res Commun. 2006 Jun 9;344(3):780-5. doi: 10.1016/j.bbrc.2006.03.197. Epub 2006 Apr 17. PMID 16631114
- [Background] Sung JK, Koh JH, Lee MY, Kim BH, Nam SM, Kim JH, Yoo JH, Kim SH, Hong SW, Lee EY, Choi R, Chung CH. Aldose reductase inhibitor ameliorates renal vascular endothelial growth factor expression in streptozotocin-induced diabetic rats. Yonsei Med J. 2010 May;51(3):385-91. doi: 10.3349/ymj.2010.51.3.385. PMID 20376891
- [Background] Sawada O, Kawamura H, Kakinoki M, Sawada T, Ohji M. Vascular endothelial growth factor in the aqueous humour in eyes with myopic choroidal neovascularization. Acta Ophthalmol. 2011 Aug;89(5):459-62. doi: 10.1111/j.1755-3768.2009.01717.x. Epub 2010 Jan 22. PMID 20102348
- [Background] Gao G, Li Y, Zhang D, Gee S, Crosson C, Ma J. Unbalanced expression of VEGF and PEDF in ischemia-induced retinal neovascularization. FEBS Lett. 2001 Feb 2;489(2-3):270-6. doi: 10.1016/s0014-5793(01)02110-x. PMID 11165263
- [Background] Kwak N, Okamoto N, Wood JM, Campochiaro PA. VEGF is major stimulator in model of choroidal neovascularization. Invest Ophthalmol Vis Sci. 2000 Sep;41(10):3158-64. PMID 10967078
- [Background] Okamura N, Ito Y, Shibata MA, Ikeda T, Otsuki Y. Fas-mediated apoptosis in human lens epithelial cells of cataracts associated with diabetic retinopathy. Med Electron Microsc. 2002 Dec;35(4):234-41. doi: 10.1007/s007950200027. PMID 12658358
- [Background] Kim B, Kim SY, Chung SK. Changes in apoptosis factors in lens epithelial cells of cataract patients with diabetes mellitus. J Cataract Refract Surg. 2012 Aug;38(8):1376-81. doi: 10.1016/j.jcrs.2012.04.026. Epub 2012 Jun 23. PMID 22727992
- [Background] Gregory MS, Repp AC, Holhbaum AM, Saff RR, Marshak-Rothstein A, Ksander BR. Membrane Fas ligand activates innate immunity and terminates ocular immune privilege. J Immunol. 2002 Sep 1;169(5):2727-35. doi: 10.4049/jimmunol.169.5.2727. PMID 12193747
- [Background] Griffith TS, Yu X, Herndon JM, Green DR, Ferguson TA. CD95-induced apoptosis of lymphocytes in an immune privileged site induces immunological tolerance. Immunity. 1996 Jul;5(1):7-16. doi: 10.1016/s1074-7613(00)80305-2. PMID 8758890
- [Background] Sotozono C, Sano Y, Suzuki T, Tada R, Ikeda T, Nagata S, Kinoshita S. Soluble Fas ligand expression in the ocular fluids of uveitis patients. Curr Eye Res. 2000 Jan;20(1):54-7. PMID 10611715
- [Background] Roychoudhury J, Herndon JM, Yin J, Apte RS, Ferguson TA. Targeting immune privilege to prevent pathogenic neovascularization. Invest Ophthalmol Vis Sci. 2010 Jul;51(7):3560-6. doi: 10.1167/iovs.09-3890. Epub 2010 Feb 17. PMID 20164456
- [Background] Kovacic N, Grcevic D, Katavic V, Lukic IK, Marusic A. Targeting Fas in osteoresorptive disorders. Expert Opin Ther Targets. 2010 Oct;14(10):1121-34. doi: 10.1517/14728222.2010.522347. PMID 20854180
- [Background] Berkkanoglu M, Guzeloglu-Kayisli O, Kayisli UA, Selam BF, Arici A. Regulation of Fas ligand expression by vascular endothelial growth factor in endometrial stromal cells in vitro. Mol Hum Reprod. 2004 Jun;10(6):393-8. doi: 10.1093/molehr/gah060. Epub 2004 Apr 8. PMID 15073283
- [Background] Nolan A, Weiden MD, Thurston G, Gold JA. Vascular endothelial growth factor blockade reduces plasma cytokines in a murine model of polymicrobial sepsis. Inflammation. 2004 Oct;28(5):271-8. doi: 10.1007/s10753-004-6050-3. PMID 16134000
- [Background] Devaraj S, Tobias P, Jialal I. Knockout of toll-like receptor-4 attenuates the pro-inflammatory state of diabetes. Cytokine. 2011 Sep;55(3):441-5. doi: 10.1016/j.cyto.2011.03.023. Epub 2011 Apr 16. PMID 21498084
- [Background] Almeida DR, Johnson D, Hollands H, Smallman D, Baxter S, Eng KT, Kratky V, ten Hove MW, Sharma S, El-Defrawy S. Effect of prophylactic nonsteroidal antiinflammatory drugs on cystoid macular edema assessed using optical coherence tomography quantification of total macular volume after cataract surgery. J Cataract Refract Surg. 2008 Jan;34(1):64-9. doi: 10.1016/j.jcrs.2007.08.034. PMID 18165083
- [Background] Almeida DR, Khan Z, Xing L, Bakar SN, Rahim K, Urton T, El-Defrawy SR. Prophylactic nepafenac and ketorolac versus placebo in preventing postoperative macular edema after uneventful phacoemulsification. J Cataract Refract Surg. 2012 Sep;38(9):1537-43. doi: 10.1016/j.jcrs.2012.04.034. Epub 2012 Jul 15. PMID 22795976